CLINICAL TRIAL: NCT06963762
Title: The Effect of Mirror Therapy Applied to Stroke Patients on Motor-Sensory Status and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, AHMET ŞİMŞEK, PhD student, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: ATAÜNİ-SBE-AS-03
Record Dates: First submitted 2025-04-10; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Mirror Movement Therapy; Rehabilitation
Keywords: stroke; mirror movement therapy; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional rehabilitation group (Experimental)
  Interventions: Behavioral: Conventional rehabilitation will be applied
- group receiving mirror therapy along with conventional rehabilitation (Experimental)
  Interventions: Behavioral: Mirror therapy will be applied along with conventional rehabilitation

INTERVENTIONS:
Behavioral: Conventional rehabilitation will be applied — Conventional rehabilitation will be applied for 30 minutes, 4 times a week for 4 weeks.
  Arms: conventional rehabilitation group
Behavioral: Mirror therapy will be applied along with conventional rehabilitation — In addition to conventional rehabilitation, patients in the experimental group will receive mirror therapy for 30 minutes, 4 times a week for 4 weeks.
  Arms: group receiving mirror therapy along with conventional rehabilitation

SUMMARY:
Purpose: The research will be conducted to evaluate the effect of Mirror Therapy applied to Stroke Patients on motor-sensory status and quality of life.

Method: The research will be carried out as a randomized controlled experimental study at Bilecik Training and Research Hospital and Bozüyük State Hospital between 01.08.2024-01.05.2025. The population of the research consists of 350 people. Individuals will be distributed to the experimental (30) and control (30) groups by simple randomization method. In collecting research data; The patient introduction form, Brunnstrom Staging and SF-36 Quality of Life Scale will be administered to the patients in both groups by the researcher using face-to-face interview technique (pre-test). Patients in the experimental group will be informed about mirror therapy.

In addition to conventional rehabilitation, patients in the experimental group will receive mirror therapy for 30 minutes, 4 times a week for 4 weeks.

Patients in the control group will only receive conventional rehabilitation for 30 minutes, 4 times a week for 4 weeks. At the end of the 4th week, patients in both groups will be administered Brunnstrom Staging and SF-36 Quality of Life Scale (posttest).

If both groups are discharged before 4 weeks, the planned practices will continue at home.

ELIGIBILITY:
Inclusion Criteria:

1. Being literate,
2. Being over the age of 18,
3. Having sufficient communication skills to answer oral and written questions and follow instructions,
4. Having been diagnosed with a stroke and at least 6 days have passed since it occurred,
5. Not having severe vision problems,
6. Not having a vertigo problem,
7. Not having been diagnosed with epilepsy,
8. Upper extremity Stage 2 and above in Brunnstrom staging
9. Lower extremity Stage 2 and above in Brunnstrom staging

Exclusion Criteria:

1. Being under 18 years of age
2. Upper extremity Stage 2 and below in Brunnstrom staging
3. In Brunnstrom staging, Lower extremity Stage 2 and below

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Brunnstrom Motor-Sensory Staging | 1 month
  Brunnstrom staging, which divides the motor recovery process in hemiplegic patients into 6 periods, was used in the upper extremity motor-sensory evaluation of the patients. Brunnstrom staging; Reveals the stages of recovery of patients from hemiplegia after a stroke. It was developed by Swedish physiatrist Signe Brunnström and highlights the synergistic pattern that develops during recovery from stroke.

SECONDARY OUTCOMES:
SF-36 Quality of Life Scale | 1 month
  The SF-36 quality of life scale was used to determine the patients' quality of life. The scale was developed by Ware and Sherbourne in 1992. The validity and reliability of the scale in Turkish was conducted by Koçyiğit. Quality of life scale; It contains 36 statements evaluating 2 main dimensions and 8 sub-dimensions. The scale has Likert type scoring. 35 of the 36 statements in the scale are evaluated considering the last 4 weeks.